CLINICAL TRIAL: NCT02214212
Title: TWILIGHT: Effect of Light Exposure During Acute Rehabilitation on Sleep After TBI.
Brief Title: TWILIGHT Study: Effect of Light Exposure During Acute Rehabilitation on Sleep After TBI
Acronym: TWILIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); University of North Texas Health Science Center (Other)
Responsible Party: Principal Investigator, Jeanne Hoffman, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00000219
Record Dates: First submitted 2014-07-31; First posted 2014-08-12 (Estimated); Results first posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Traumatic Brain Injury; TBI; Sleep
Keywords: traumatic brain injury; TBI; Sleep; Bright White Light Therapy; Red Light Therapy; Recovery; Central Nervous System Diseases; Brain Diseases; Nervous System Diseases; Signs and Symptoms; Rehabilitation; Actigraphy
MeSH Terms: conditions — Brain Injuries, Traumatic; Central Nervous System Diseases; Brain Diseases; Nervous System Diseases; Signs and Symptoms | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Red Light (RL) (Active Comparator): Intervention/Device:
  This patient group will receive 30 minutes of red light daily for a period of 10 days in the morning. Identical baseline and outcome testing will be completed for both arms.
  Interventions: Device: Red Light (RL)
- Bright White Light (BWL) (Experimental): Intervention/Device:
  This patient group will receive 30 minutes of bright white light daily for a period of 10 days in the morning. Identical baseline and outcome testing will be completed for both arms.
  Interventions: Device: Bright White Light (BWL)

INTERVENTIONS:
Device: Bright White Light (BWL) — The device emitting BWL will be placed 24 inches from the participant's face on a pre-measured table. The participant will spend 30 minutes with the eyes open in front of the device. This will occur each morning for 10 days.
  Other Names: Litebook® (Bright White Light)
  Arms: Bright White Light (BWL)
Device: Red Light (RL) — The device emitting RL will be placed 24 inches from the participant's face on a pre-measured table. The participant will spend 30 minutes with the eyes open in front of the device. This will occur each morning for 10 days.
  Other Names: Litebook® (Red Light)
  Arms: Red Light (RL)

SUMMARY:
This study proposes to investigate how well Bright White Light Therapy will work in the acute inpatient rehabilitation units for people whom have experienced a traumatic brain injury for the purpose of treating sleep disruption. Participants will be assessed based on sleep efficiency, thinking abilities, therapy participation, and perception of fatigue/sleepiness. In previous studies dim red light has not had the same effects on function as bright white light, and will be chosen for use as a placebo. Each subject will be randomized to receive 30 minutes of either Bright White Light Therapy or Red Light Treatment each morning for 10 days.

To measure the effect of this treatment, the investigators will measure the each participants sleep daily by using an actigraph watch. This watch will record movement continuously. The investigators will also measure the subjects' report of how well they slept, whether fatigue is present, and how attentive they are before and after treatment.

Research Hypothesis:

In persons with TBI, prospectively compare overnight sleep in a cohort exposed to morning Bright White Light with a comparison group exposed to Red Light in an acute inpatient rehabilitation setting.

DETAILED DESCRIPTION:
The investigators will recruit persons with moderate to severe traumatic brain injury (TBI) on admission to intensive rehabilitation units. Consented participants (who meet all inclusion and exclusion criteria) will wear an actigraphy watch for 2 nights to obtain a baseline for sleep pattern identification. Prior to treatment, baseline measures (detailed below) will be obtained. Participants will be randomized to receive either Bright White Light (BWL) or Red Light (RL) treatment. Light therapy treatments will be given for 30 minutes daily in the morning for 10 days, and an Actiwatch will be worn continuously during that period. At the end of 10 days, outcome measures will be obtained (as below). The specific period of treatment may be affected by the length of stay on the rehabilitation unit. For lengths of stay less than the 10 days, subjects will receive the intervention until the day of discharge at which time the outcome measures will be administered. The investigators primary outcome measure with be the actigraphic measurement of sleep efficiency. Other secondary measures will be participation in therapy, sleepiness, and attention. The investigators will also evaluate the anticipated device costs and clinical staff burden involved in utilizing light therapy exposure in an inpatient rehabilitation clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Have experienced a moderate to severe TBI.

Defined by any of the following:

1. Loss of Consciousness greater than 30 minutes.
2. Emergency Room admission with a Glasgow Coma Scale of 12 or below.
3. Intracranial abnormalities on imaging.
4. Post-traumatic amnesia that lasts more than 24 hours.

   * Admitted to acute inpatient rehabilitation unit at Harborview Medical Center within 3 months of their Traumatic Brain Injury.
   * Able to communicate in English.
   * Between the ages of 18 and 70 years old
   * Have a clinician rating of the presence of a sleep disturbance (using the Makley scale)
   * Have some vision in one or both eyes.
   * Have a Body Mass Index lower than 40 kg/m2

Exclusion Criteria:

Unable to enroll if any of the following are true

* Complete blindness
* Absence of eye opening or disorders of consciousness (Rancho level 1-3).
* Tetraplegia with less than antigravity strength in all myotomes caudal to C6 level given the limitations on measuring movements with actigraphy in this population (i.e. cannot reliably detect upper extremity or lower extremity movement with this level of paralysis).
* Past medical history of retinal pathology
* Past medical history of light sensitivity
* Past medical history of narcolepsy
* Past medical history of bipolar disorder
* Past medical history of obstructive sleep apnea
* Suspected sleep apnea. (Determined by administering the Berlin questionnaire)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne M Hoffman, PhD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bell KR, Fogelberg D, Barber J, Nakase-Richardson R, Zumsteg JM, Dubiel R, Dams-O'Connor K, Hoffman JM. The effect of phototherapy on sleep during acute rehabilitation after traumatic brain injury: a randomized controlled trial. Brain Inj. 2021 Jan 18;35(2):180-188. doi: 10.1080/02699052.2021.1871952. Epub 2021 Jan 17. PMID 33459040

RESULTS

PARTICIPANT FLOW:
Groups:
- Red Light (RL): Intervention/Device:
  This patient group will receive 30 minutes of red light daily for a period of 10 days in the morning. Identical baseline and outcome testing will be completed for both arms.
  Red Light (RL): The device emitting RL will be placed 24 inches from the participant's face on a pre-measured table. The participant will spend 30 minutes with the eyes open in front of the device. This will occur each morning for 10 days.
- Bright White Light (BWL): Intervention/Device:
  This patient group will receive 30 minutes of bright white light daily for a period of 10 days in the morning. Identical baseline and outcome testing will be completed for both arms.
  Bright White Light (BWL): The device emitting BWL will be placed 24 inches from the participant's face on a pre-measured table. The participant will spend 30 minutes with the eyes open in front of the device. This will occur each morning for 10 days.
Period: Overall Study
Arm/Group | Red Light (RL) | Bright White Light (BWL)
Started | 66 | 65
Completed | 57 | 59
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Red Light (RL) | Bright White Light (BWL) | Total
Number analyzed (Participants) | 66 | 65 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (2.7) | 39.8 (2.6) | 41 (2.7)
Age, Customized [Count of Participants; unit: Participants]
  <25 | 15 | 12 | 27
  25-39 | 15 | 24 | 39
  40-54 | 19 | 15 | 34
  55+ | 17 | 12 | 29
  Unknown | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 44 | 46 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 43 | 48 | 91
  Black | 10 | 6 | 16
  Asian/Pacific Islander | 2 | 0 | 2
  Native American | 4 | 2 | 6
  Hispanic | 5 | 7 | 12
  Other | 2 | 0 | 2
  Unknown | 0 | 2 | 2
Education [Mean (Standard Deviation); unit: years] | 13 (2.3) | 14 (2.5) | 13.5 (2.5)
Marital Status [Number; unit: participants]
  Single | 24 | 27 | 51
  Married | 25 | 25 | 50
  Div/Sep/Widow | 16 | 11 | 27
  Unknown | 1 | 2 | 3
Cause of Injury [Number; unit: Participants]
  Vehicular | 28 | 42 | 70
  Violence | 11 | 3 | 14
  Fall | 17 | 13 | 30
  Pedestrian | 3 | 6 | 9
  Other | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Actigraphy Data
Description: Sleep efficiency scores derived from actigraphy data will be the primary outcome. We will set the Actiwatch to record activity data in 60-second intervals. Actigraphy data will be automatically scored with Actiware software (Respironics, Philips Healthcare), which uses validated algorithms to determine whether an epoch of activity is "sleep" or "wake" (Cole RJ, 1992). Typically there is a lack of a consistent sleep/wake cycle in the study population, therefore we will be using sleep efficiency and total sleep time scores obtained during a set night-time interval (2200 to 0600) as the primary index of sleep function, as has been used in previous publications[39, 40]. We will be comparing average between group differences between the BWL and RL groups at baseline and after 10 days of light therapy.
Time Frame: Average percent sleep efficiency (0-100) at baseline and after 10 days of light exposure
Population: Of the overall enrollment number of 131 participants, we were able to obtain completed data for this measure on 117 (or 89%) and a breakdown between groups for light exposure of 57=Red Light and 60=Bright White Light.
Measure: Mean (Standard Deviation); unit: percentage of sleep efficiency (0-100)
Groups:
- Red Light (RL): The Red Light group was exposed to RL (control) for 30 minutes each morning between 0730 and 0930 for up to 10 days. Both interventions were delivered using a Litebook® with visually identical cases.
- Bright White Light (BWL): The intervention group was exposed to BWL (active treatment) for 30 minutes each morning between 0730 and 0930 for up to 10 days. Both interventions were delivered using a Litebook® with visually identical cases.
Arm/Group | Red Light (RL) | Bright White Light (BWL)
Number analyzed (Participants) | 57 | 60
percentage of sleep efficiency (0-100)
  Baseline | 72 (17) | 76 (17)
  After 10 days of light exposure | 76 (11) | 77 (13)
Statistical Analysis 1: Comparison: Red Light (RL) vs Bright White Light (BWL); Test type: Superiority; p = .955, Mixed Models Analysis; Mixed-effects model used an unstructured correlation matrix, adjusting for treatment, time (linear) and the interaction as fixed effects; Slope = -0.16, 95% CI 2-sided [-5.69 to 5.37] — The reported effect size has been expressed as the modelled difference in sleep efficiency improvement from day 1 to day 10. A positive effect size indicates a higher score in the white-light arm

2. Secondary Outcome: Barrow Neurological Institute Fatigue Scale (BNI-FS)
Description: The Barrow Neurological Institute Fatigue Scale (BNI-FS; Fatigue Outcome) is an 11-point scale that examines fatigue during acute recovery from TBI. Scores on items 1-10 may range from 1 (rarely a problem), 2-3 (occasional problem but not frequent), 4-5 (a frequent problem), 6-7 (a problem most of the time). The last item is a general rating of fatigue from 0 (not a problem) to 10 (a severe problem). The total BNI-FS is a sum of the first 10 items (0-70), where higher scores indicate worse outcome.
  The BNI-FS is a scale that was designed to examine fatigue during acute recovery from TBI. The clinical staff involved in the care of these subjects were asked to rate the phototherapy intervention for ease of use, perceived relevance to rehabilitation care, and impression of effectiveness.
Time Frame: At Baseline and After 10 Days of Light Exposure
Population: Statistical significance by mixed-effects regression adjusting for site, FIM admit cognitive, FIM admit motor. (Incident and education did not improve any of the models.) Of the overall enrollment number of 131 participants, we were able to obtain completed data for this measure on 116 (or 88%).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Red Light (RL): The Red Light group was exposed to RL (comparator) for 30 minutes each morning between 0730 and 0930 for up to 10 days. Both interventions were delivered using a Litebook® with visually identical cases.
Arm/Group | Red Light (RL) | Bright White Light (BWL)
Number analyzed (Participants) | 55 | 61
score on a scale
  Baseline | 23.7 (15.6) | 26.5 (14.0)
  After 10 days of light exposure | 15.6 (13.0) | 18.3 (16.3)
Statistical Analysis 1: Comparison: Red Light (RL) vs Bright White Light (BWL); Test type: Superiority; p = .807, Mixed Models Analysis; Mean Difference (Net) = 0.69, 95% CI 2-sided [-4.90 to 6.29]

3. Secondary Outcome: Functional Independence Measure (FIM) - Motor
Description: Functional Independence Measure (FIM) is the most widely accepted functional assessment measure in use in the rehabilitation community. The FIM is an 18-item ordinal scale, used with all diagnoses within a rehabilitation population. Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item. Motor subscale (the sum of the individual motor subscale items) will be a value between 13 and 91.
Time Frame: Administered at baseline (admission to unit) and after Day 10 of intervention (or at the day of discharge from the rehabilitation unit)
Population: Of the overall enrollment number of 131 participants, we were able to obtain completed data for this measure on 124 (or 95%). The Functional Independence Measure (FIM) was completed at Rehab Admit and again at Rehab Discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Red Light (RL) | Bright White Light (BWL)
Number analyzed (Participants) | 62 | 62
score on a scale
  FIM Motor -Rehab Admit | 36.5 (18.9) | 38.5 (17.3)
  FIM Motor - Rehab Discharge | 68.2 (16.0) | 69.8 (12.8)
Statistical Analysis 1: Comparison: Red Light (RL) vs Bright White Light (BWL); Test type: Superiority; p = .847, Mixed Models Analysis; Mixed-effects model adjusts for treatment, time (pre/post), site, FIM admit cognitive/motor, and the treatment/time as fixed effects; Mean Difference (Net) = -0.48, 95% CI 2-sided [-5.38 to 4.43]

4. Secondary Outcome: Symbol Digit Modalities Test
Description: The Symbol Digit Modalities Test (SDMT) is a pencil and paper test for attention that takes approximately five minutes to administer and is frequently used in evaluations after TBI. The SDMT was administered at enrollment and after intervention. The Interagency Workgroup on TBI Outcomes selected the SDMT as CORE common data elements in TBI outcomes research. The SDMT measures attention and speed of processing (the test-taker substitutes a number for random presentations of geometric figures). Scoring involves summing the number of correct substitutions within the 90 second interval (min=0, max = 110), with higher scores representing better attention/speed of processing.
Time Frame: Administered at Baseline and After 10 Days of Light Exposure
Population: Of the overall enrollment number of 131 participants, we were able to obtain completed data for this measure on 79 participants (or 60%).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Red Light (RL) | Bright White Light (BWL)
Number analyzed (Participants) | 39 | 40
score on a scale
  Baseline | 21.3 (13.3) | 21.6 (12.3)
  After 10 days light exposure | 25.9 (14.4) | 29.0 (12.0)
Statistical Analysis 1: Comparison: Red Light (RL) vs Bright White Light (BWL); Test type: Superiority; p = .252, Mixed Models Analysis; Statistical significance by mixed-effects regression adjusts for time (pre/post), site, FIM admit cognitive, FIM admit motor as fixed effects; Mean Difference (Net) = 3.14, 95% CI 2-sided [-2.29 to 8.56]

5. Secondary Outcome: Positive and Negative Affect Schedule - Positive
Description: The Positive and Negative Affect Schedule (PANAS; Mood Outcome) includes a total of 20 items of affect with 10 focused on positive affect and 10 focused on negative affect. The total score of the PANAS: Positive is the sum of the 10 positive items which are rated on a likert scale ranging from 1=very slightly or not at all to 5=extremely. For the total positive score, a higher score indicates more positive affect. affect. Scores can range from 10-50 for Positive Affect.
Time Frame: Administered at Baseline and After 10 Days of Light Exposure
Population: Of the overall enrollment number of 131, we were able to obtain completed data for this measure on 118 participants (or 90%).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Red Light (RL): This group was exposed to Red Light (RL) (control) for 30 minutes each morning between 0730 and 0930 for up to 10 days. Both interventions were delivered using a Litebook® with visually identical cases.
- Bright White Light (BWL): This group was exposed to BWL (active treatment) for 30 minutes each morning between 0730 and 0930 for up to 10 days. Both interventions were delivered using a Litebook® with visually identical cases.
Arm/Group | Red Light (RL) | Bright White Light (BWL)
Number analyzed (Participants) | 57 | 61
score on a scale
  Baseline | 31.8 (9.0) | 30.9 (9.3)
  After 10 Days of Light Exposure | 34.0 (8.8) | 34.2 (9.0)
Statistical Analysis 1: Comparison: Red Light (RL) vs Bright White Light (BWL); Test type: Superiority; p = .722, Mixed Models Analysis; Mean Difference (Net) = 0.67, 95% CI 2-sided [-3.08 to 4.4]

6. Secondary Outcome: Positive and Negative Affect Schedule - Negative
Description: The Positive and Negative Affect Schedule (PANAS; Mood Outcome) includes a total of 20 items of affect with 10 focused on positive affect and 10 focused on negative affect. The total score of the PANAS: Negative is the sum of the 10 negative items which are rated on a likert scale ranging from 1=very slightly or not at all to 5=extremely. For the total negative score, a higher score indicates more negative affect. affect. Scores can range from 10-50 for Negative Affect.
Time Frame: Administered at baseline and after 10 days of light exposure
Population: Of the overall enrollment number of 131, we were able to obtain completed data for this measure on 119 participants (or 91%).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Red Light (RL) | Bright White Light (BWL)
Number analyzed (Participants) | 58 | 61
score on a scale
  Baseline | 19.7 (8.7) | 19.6 (8.2)
  After 10 days of light exposure | 18.4 (8.6) | 17.1 (7.2)
Statistical Analysis 1: Comparison: Red Light (RL) vs Bright White Light (BWL); Test type: Superiority; p = .253, Mixed Models Analysis; Mean Difference (Net) = -2.25, 95% CI 2-sided [-6.13 to 1.64]

7. Secondary Outcome: Karolinska Sleepiness Scale (KSS)
Description: The Karolinska Sleepiness Scale (KSS; Sleepiness Outcome) is a single-question with a 9-point Likert scale (1 = extremely alert, 9 = extremely sleepy, fighting sleep) measuring subjective sleepiness at the time of report.
Time Frame: Administered at Baseline and after 10 Days of Light Exposure
Population: Of the overall enrollment number of 131, we were able to obtain completed data for this measure on 121 participants (or 92%).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Red Light (RL) | Bright White Light (BWL)
Number analyzed (Participants) | 59 | 62
score on a scale
  Baseline | 4.1 (1.8) | 4.1 (1.8)
  After 10 Days of Light Exposure | 4.1 (2.0) | 3.7 (1.7)
Statistical Analysis 1: Comparison: Red Light (RL) vs Bright White Light (BWL); Test type: Superiority; p = .351, Mixed Models Analysis; [statistical method as in outcome 3, analysis 1]; Mean Difference (Net) = -0.39, 95% CI 2-sided [-1.21 to 0.44] — A positive effect size indicates a higher score in the bright white light (BWL) intervention arm

8. Secondary Outcome: Makley Scale
Description: The Makley scale is a 4-point ordinal scale which allows staff to score sleep as follows:
  0 = asleep; 1 = drowsy/falling asleep; 2 = drowsy/waking up; 3 = awake.
Time Frame: A sleep log was completed every 2 hours during the night (2200 until 0600) on each patient by the unit nursing staff hours for 12 nights or until discharge from the hospital (2 nights baseline and after 10 nights of intervention light exposure)
Population: 1:1 comparison; Of the overall enrollment number of 131, we were able to obtain completed data for this measure on 117 participants (or 89%).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Red Light (RL) | Bright White Light (BWL)
Number analyzed (Participants) | 57 | 60
score on a scale
  Baseline | 0.58 (0.38) | 0.67 (0.54)
  After 10 Days of Light Exposure | 0.59 (0.29) | 0.61 (0.33)
Statistical Analysis 1: Comparison: Red Light (RL) vs Bright White Light (BWL); Test type: Superiority; p = .910, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Slope = 0.00, 95% CI 2-sided [-0.03 to 0.03] — The reported effect size has been expressed as the modelled difference in the Makley scale score improvement from day 1 to day 10. A positive effect size indicates a higher score in the white-light arm

9. Secondary Outcome: Functional Independence Measure (FIM) - Cognitive
Description: Functional Independence Measure (FIM) is the most widely accepted functional assessment measure in use in the rehabilitation community. The FIM is an 18-item ordinal scale, used with all diagnoses within a rehabilitation population. Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item. Cognition subscale (the sum of the individual cognition subscale items) will be a value between 5 and 35.
Time Frame: Administered at baseline (admission to unit) and after Day 10 of light exposure (or at the day of discharge from the rehabilitation unit)
Population: Of the overall enrollment number of 131, we were able to obtain completed data for this measure on 124 participants (or 95%).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Red Light (RL) | Bright White Light (BWL)
Number analyzed (Participants) | 62 | 62
score on a scale
  FIM Cognitive- Admit | 15.1 (6.9) | 14.3 (6.3)
  FIM Cognitive-Discharge | 24.7 (5.7) | 24.1 (5.1)
Statistical Analysis 1: Comparison: Red Light (RL) vs Bright White Light (BWL); Test type: Superiority; p = 0.19, Mixed Models Analysis; Mixed-effects model adjusts for treatment time (pre/post); Mean Difference (Net) = .857, 95% CI 2-sided [-1.93 to 2.32]

10. Other Pre Specified Outcome: Cooperation Measure (Therapy Outcome)
Description: Cooperation Measure (Therapy Outcome). Patient cooperation was rated using a visual analogue scale (VAS) ranging from 0%-not cooperative to 100%- fully cooperative.10 Staff physical therapists were asked to rate cooperation both prior to initiation and after completion of phototherapy.
Time Frame: Collected at Baseline and after 10 days of light exposure
Population: Of the overall enrollment number of 131, we were able to obtain completed data for this measure on 123 participants (or 94%).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Red Light (RL) | Bright White Light (BWL)
Number analyzed (Participants) | 60 | 63
score on a scale
  Baseline | 77.3 (27.3) | 84.5 (22.5)
  After 10 Days of Light Exposure | 86.6 (23.0) | 89.4 (22.5)
Statistical Analysis 1: Comparison: Red Light (RL) vs Bright White Light (BWL); Test type: Superiority; p = .345, Mixed Models Analysis; Mixed-effects model adjusts for treatment, time (pre/post), FIM admit cognitive, site, FIM admit motor as mixed effects; Mean Difference (Net) = -4.80, 95% CI 2-sided [-14.83 to 5.24]

ADVERSE EVENTS:
Time Frame: Adverse Event Reporting Period The study period during which adverse events were reported was the period from the initiation of study procedures to the end of the study treatment follow-up. For this study, the study treatment follow-up was 2 days following the last study treatment (Day 15).
Arm/Group | Red Light (RL) | Bright White Light (BWL)
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/65
Other Adverse Events (participants affected / at risk) | 0/66 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT02214212/Prot_SAP_000.pdf